CLINICAL TRIAL: NCT02515201
Title: Heparin Versus Taurolidine to Bloodstream Infection Prevention Related in Central Venous Catheter in Children With Intestinal Failure
Brief Title: Heparin Versus Taurolidine to Bloodstream Infection Prevention Related in Central Venous Catheter in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Helena Ayako Sueno Goldani, Helena Goldani, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 140291
Record Dates: First submitted 2015-07-19; First posted 2015-08-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections | interventions — taurolidine; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taurolidine (Active Comparator): Taurolidine be held in each infusion central venous catheter lumen with a volume that varies in accordance with the lumen via the catheter. The solution will be administered every day while the patient is on break from parenteral nutrition, and the catheter solution residence time will be the same time of the break from parenteral nutrition. Taurolidine infusion will be used TaurolockTM with ampoule presentation containing 3 ml.
  Interventions: Drug: Taurolidine
- Heparin (Active Comparator): Heparin be held in each infusion central venous catheter lumen with a volume that varies in accordance with the lumen via the catheter. The solution will be administered every day while the patient is on break from parenteral nutrition, and the catheter solution residence time will be the same time of the break from parenteral nutrition. Heparin infusion will be used with heparin solution contain 50 International Unit (UI)/ml.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Taurolidine — taurolidine in central catheter lumen
  Other Names: Taurolock
  Arms: Taurolidine
Drug: Heparin — heparin in central venous catheter lumen
  Other Names: heparin solution
  Arms: Heparin

SUMMARY:
Clinical trial, that aim is evaluation of the use of taurolidine and heparin in the prevention of bloodstream infection in venous catheter in children with intestinal failure.

DETAILED DESCRIPTION:
Will be collected data about sociodemographics : date of birth, hospitalization and which is use (taurolidine or heparin), sex, underlying disease and associated co-morbidities.

About central venous catheter will be collect: catheter type in each period, the number of lumens, date of insertion of each catheter usage time, reason for removal of the catheter insertion site and catheter material (silicone or polyurethane ).

Data relating to parenteral nutrition will also be collected: osmolarity of parenteral nutrition, infusion time every 24 hours and concentration of glucose parenteral nutrition bag.

It will be used for aseptic handling technique of the solutions, as well as for handling the connections of the central catheter. For preparation and administration of taurolidine and heparin is used an operations manual that was made for the authors. Patients are divided into two groups: taurolidine or heparin.

ELIGIBILITY:
Inclusion Criteria:

* The population will consist of patients 30 days of life to fourteen years old, admitted to the pediatric inpatient units, with intestinal failure receiving parenteral nutrition through a central venous catheter and at least eight weeks of use forecast.

Exclusion Criteria:

* Children will be excluded other associated diseases that occur with frequent use of antibiotics, for example, cystic fibrosis, primary or acquired immunodeficiency. Also excluded are the children admitted that they are not accompanied by a responsible family recognition, or accompanied by responsible under the age of 18 years. Children with allergic reactions to the use of some of the solutions (taurolidine or heparin) will be suspended medication and receive appropriate treatment. Although these children have stopped the use of medication, will be followed according to the assessment protocol by the end of the study.

Ages: 30 Days to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Bloodstream infection related to the use of central venous catheter | 1 year
  Bloodstream infection related to the use of central venous catheter is defined as positive culture of microorganisms in blood samples collected from the central venous catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carolina Witkowski, MD, Study Chair — Hospitall de Clínicas de Porto Alegre; Adriano Taniguchi, MD, Study Chair — Hospital de Clínicas de Porto Alegre; Elza Mello, PhD, Study Chair — Hospital de Clínicas de Porto Alegre; Suzi Camey, PhD, Study Chair — Hospital de Clínicas de Porto Alegre; Helena Goldani, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre